CLINICAL TRIAL: NCT05316376
Title: Effect of Albumin-bound Paclitaxel Plus Carboplatin Compared With Paclitaxel Plus Carboplatin in Patients Receiving Neoadjuvant Chemotherapy for Advanced Ovarian, Fallopian Tube or Peritoneal Cancer: A Phase 2 Single Center Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-KY-036
Record Dates: First submitted 2022-03-31; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Albumin-Bound Paclitaxel; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Dd-nab-paclitaxel (100 mg/m2, days 1, 8, and 15, every 4 weeks), combined with carboplatin (AUC = 5, days 1), dd-nab TC regimen every 4 weeks will be given to the patients in study group, while for the patients in control group, paclitaxel (175 mg/m2, day 1) combined with carboplatin (AUC=6, day1) will administered.
Who Masked: Investigator
Masking Description: Pathological slides of omentum will be independently reviewed by two pathologists who will be blinded to the randomization to determine the CRS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dd-nabTC (Experimental): albumin-bound paclitaxel (100 mg/m2, days 1, 8, and 15, every 4 weeks) combined with carboplatin (AUC = 5, day 1, every 4 weeks)
  Interventions: Drug: albumin-bound paclitaxel
- CONTROL (Active Comparator): paclitaxel (175 mg/m2, day 1, every 4 weeks) combined with carboplatin (AUC=6, day1, every 4 weeks)
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: albumin-bound paclitaxel — albumin-bound paclitaxel (100 mg/m2, days 1, 8, and 15, every 4 weeks) combined with carboplatin (AUC = 5 day 1, every 4 weeks)
  Arms: dd-nabTC
Drug: paclitaxel — paclitaxel (175 mg/m2, day 1, every 3 weeks) combined with carboplatin (AUC=6, day1, every 3 weeks)
  Arms: CONTROL

SUMMARY:
Neoadjuvant chemotherapy (NACT) is an important option for patients with advanced ovarian cancer. Paclitaxel plus carboplatin is the first-line regimen for ovarian cancer NACT patients. However, the efficacy of NACT is controversial, how to improve the efficacy become an urgent problem to be solved in the treatment of ovarian cancer. It has been confirmed that the dose-intensive paclitaxel combined carboplatin regimen can improve the prognosis in Asian patients with advanced ovarian cancer. However, this protocol has a low rate of complete tumor remission after NACT (4%) with toxicities and high probability of severe hypersensitivity reactions. Albumin-bound paclitaxel has the characteristics of tumor targeting, low allergenicity. We propose that dose-dense albumin-bound paclitaxel (ddnab-paclitaxel) (100 mg/m2, days 1, 8, and 15) combined with carboplatin (AUC = 5 days 1, 4 weeks) regimen may be superior to the paclitaxel plus carboplatin regimen. We conducted this Phase II randomized controlled study to testify the efficacy of dd-nab paclitaxel. 57 stage IIIC-IV patients with high-grade epithelial, fallopian tube, and peritoneal cancer who are unable to undergo optimal cytoreduction and receive NACT after tumor biopsy will be recruited. The regimen for the study group is albumin-bound paclitaxel (100 mg/m2, days 1, 8, and 15 doses) combined with carboplatin (AUC = 5 day 1, 4 weeks), while patients in the control group use paclitaxel (175 mg/m2, day 1) combined with carboplatin (AUC=6, day1). Interval debulking surgery(IDS) will be performed within 3-4 weeks after 3 cycles of NACT. The primary endpoint is the proportion of Chemotherapy Response Score (CRS) of 3 according to the CRS system. The secondary endpoints are progression-free survival(PFS), overall survival(OS) and the rates of complete resection and adverse events(AEs).

ELIGIBILITY:
Inclusion Criteria:

* International Federation of Gynecology and Obstetrics(FIGO) stage IIIC-IVA, HGSOC Patients with Fagotti score ≥8
* Adequate kidney function (blood creatinine 58-96 µmol/L)
* Adequate haematological function (haemoglobin ≥110g/L, leucocytes ≥4.0×109/L, neutrophils ≥2.0×109/L, platelets≥100×109/L)
* Adequate liver function (serum total bilirubin 3.4-22.2µmol/L, alanine aminotransferase (ALT) 7-40U/L, aspartate aminotransferase (AST) 13-35U/L, AST/ALT ≤1.5)
* World Health Organization(WHO) score 0-2
* expected lifespan>12 weeks

Exclusion Criteria:

* Patients who had received chemotherapy, radiotherapy or any kind of targeted therapy
* Complicated with any other known malignancies
* Patients with poor cardiopulmonary function, which would limit compliance with study requirements

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
chemotherapy response score(CRS) 3 | At the end of cycle 3 NACT (each cycle is 21 days)
  the proportion of chemotherapy response score 3

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression, assessed up to 3 years
  progression-free survival
OS | From date of randomization until the time of death from any cause, assessed up to 3 years
  overall survival
AEs | during the treatment procedure
  adverse effects of chemotherapy

IPD SHARING:
Plan to Share IPD: No